CLINICAL TRIAL: NCT03934957
Title: A Single Center, Prospective, Epidemiologic Cohort Study With Emphasis on Imaging to Improve the Identification of Individuals at Risk for Major Chronic Diseases and to Improve Early Diagnosis and Survival
Brief Title: Hamburg City Health Study - a German Cohort Study
Acronym: HCHS
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Universitäres Herzzentrum Hamburg-Eppendorf (Unknown); Martini-Klinik am UKE GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: PV5131
Record Dates: First submitted 2019-01-04; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Coronary Heart Disease; Stroke; Dementia; Cancer; Health Care; Vascular Diseases; Periodontal Diseases; Ocular Diseases; Respiratory Disease; Obesity
Keywords: Epidemiology; prospective cohort study; Nutrition; prevention; psychiatric and psychosomatic disorders
MeSH Terms: conditions — Coronary Disease; Stroke; Dementia; Neoplasms; Vascular Diseases; Periodontal Diseases; Respiration Disorders; Obesity; Psychophysiologic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma (EDTA, citrate), genomic deoxyribonucleic acid (DNA), ribonucleic acid (RNA) from whole blood and peripheral blood mononuclear cells (PBMCs), blood cells (erythrocytes, PBMCs), urine, saliva, tooth fluid, tonsils swabs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Hamburg City Health Study (HCHS) is a large, prospective, long-term, population-based cohort study and a unique research platform and network to obtain substantial knowledge about several risk and prognostic factors in major chronic diseases.

DETAILED DESCRIPTION:
A random sample of 45.000 participants between 45 and 74 years of age from the general population of Hamburg, Germany, will take part in an extensive baseline assessment at a dedicated study center. Participants undergo 13 validated and 5 novel examinations primarily targeting cardiac, arterio-venous and cerebral function and structure including extensive imaging examinations. The protocol includes self-ratings of life style and environmental conditions, , dietary habits, physical activity, professional life, psychosocial context, , digital media use, medical and family history as well as health care utilization patterns. The assessment is completed by genomic and proteomic characterization. Beyond the identification of classical risk factors for major chronic diseases and survivorship, the core intention is to develop complex models predicting health outcomes based on a multitude of examination data, imaging data and behavioral assessments. Participants at risk for coronary artery disease, atrial fibrillation, heart failure, stroke and dementia will be invited for a visit to conduct additional MRI examination either of heart or brain. Endpoint assessment of the overall sample will be completed through repeated follow-up examinations and data from involved health and pension insurances.

ELIGIBILITY:
Inclusion Criteria:

* Inhabitant of the city of Hamburg at the time of inclusion into the study (Inclusion is time of written consent)
* Age 45 to 74 years
* Personally signed informed consent

Exclusion Criteria:

* Insufficient knowledge of the German language, in order to understand study documents and computer assisted interview without translation
* Physical or psychological incapability to travel to the study center and to cooperate in the investigations

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population based cohort, participants are identified by a random sample from the official inhabitant data file divided into gender and six age strata.
Sampling Method: Probability Sample
Enrollment: 45000 (Estimated)
Dates: Start 2016-02-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
self-reported Information on changes in health in the participants | yearly up to 12 years
  coronary artery disease atrial fibrillation heart failure dementia stroke cancer such as prostate cancer and skin cancer chronic kidney diseases migraine musculoskeletal diseases such as osteoporosis and bone metastasis ocular diseases such as glaucoma, macular degeneration, fundus hypertonicus, retinal vessel disease and neoplasm oral health including periodontal disease, oropharyngeal cancer and human papillomavirus (HPV)-infection psychiatric and psychosomatic disorders such as mental disorder or late - last depression pulmonary diseases such as obstructive lung disease sexual disorder skin diseases such as psoriasis, chronic wounds and inflammation vascular diseases such as aortic aneurysm, thrombosis and peripheral arterial disease

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Blankenberg, Professor, Principal Investigator — Universitäres Herzzentrum Hamburg
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen M, Vettorazzi E, Weber P, Petersen M, Schell M, Nagele FL, Link MA, Schlemm E, Rimmele DL, Becher PM, Cheng B, Blankenberg S, Kirchhof P, Zeller T, Twerenbold R, Thomalla G. Association of Cardiac Biomarkers With Structural Brain Changes and Cognitive Impairment: Results From the Hamburg City Health Study. Neurology. 2025 Aug 12;105(3):e213865. doi: 10.1212/WNL.0000000000213865. Epub 2025 Jul 3. PMID 40609062
- [Derived] Wenzel JP, Albrecht JN, Toprak B, Petersen E, Nikorowitsch J, Cavus E, Jahnke C, Riedl KA, Adam G, Twerenbold R, Blankenberg S, Kirchhof P, Lund G, Tahir E, Mullerleile K, Radunski UK. Head-to-head comparison of cardiac magnetic resonance imaging and transthoracic echocardiography in the general population (MATCH). Clin Res Cardiol. 2025 May 12. doi: 10.1007/s00392-025-02660-1. Online ahead of print. PMID 40353872
- [Derived] Rimmele DL, Petersen EL, Affolderbach S, Petersen M, Cheng B, Mayer C, Nagele FL, Harth V, Terschuren C, Kuhn S, Zeller T, Gerloff C, Thomalla G. Differences in impact of current and former shift work on cardiovascular risk factors, carotid atherosclerosis, and white matter integrity. Sleep Adv. 2024 Jul 31;5(1):zpae056. doi: 10.1093/sleepadvances/zpae056. eCollection 2024. PMID 39156216
- [Derived] Cavus E, Schneider JN, di Carluccio E, Ziegler A, Haack A, Ojeda F, Chevalier C, Jahnke C, Riedl KA, Radunski UK, Twerenbold R, Kirchhof P, Blankenberg S, Adam G, Tahir E, Lund GK, Muellerleile K. Unrecognized myocardial scar by late-gadolinium-enhancement cardiovascular magnetic resonance: Insights from the population-based Hamburg City Health Study. J Cardiovasc Magn Reson. 2024 Summer;26(1):101008. doi: 10.1016/j.jocmr.2024.101008. Epub 2024 Feb 9. PMID 38341145
- [Derived] Rimmele DL, Borof K, Wenzel JP, Jensen M, Behrendt CA, Waldeyer C, Schnabel RB, Zeller T, Debus ES, Blankenberg S, Gerloff C, Thomalla G. Differential association of flow velocities in the carotid artery with plaques, intima media thickness and cardiac function. Atheroscler Plus. 2021 Jul 31;43:18-23. doi: 10.1016/j.athplu.2021.07.020. eCollection 2021 Sep. PMID 36644504
- [Derived] Cavus E, Schneider JN, Bei der Kellen R, di Carluccio E, Ziegler A, Tahir E, Bohnen S, Avanesov M, Radunski UK, Chevalier C, Jahnke C, Ojeda F, Kirchhof P, Blankenberg S, Adam G, Lund GK, Muellerleile K. Impact of Sex and Cardiovascular Risk Factors on Myocardial T1, Extracellular Volume Fraction, and T2 at 3 Tesla: Results From the Population-Based, Hamburg City Health Study. Circ Cardiovasc Imaging. 2022 Sep;15(9):e014158. doi: 10.1161/CIRCIMAGING.122.014158. Epub 2022 Sep 20. PMID 36126126
- [Derived] Rimmele DL, Petersen EL, Schlemm E, Kessner SS, Petersen M, Mayer C, Cheng B, Zeller T, Waldeyer C, Behrendt CA, Gerloff C, Thomalla G. Association of Carotid Plaque and Flow Velocity With White Matter Integrity in a Middle-aged to Elderly Population. Neurology. 2022 Dec 12;99(24):e2699-e2707. doi: 10.1212/WNL.0000000000201297. PMID 36123124
- [Derived] Zyriax BC, Borof K, Walter S, Augustin M, Windler E. Knowledge as to cholesterol reduction and use of phytosterol-enriched dietary foods in the general population: Insights from the Hamburg City Health Study. Atherosclerosis. 2022 Jan;341:1-6. doi: 10.1016/j.atherosclerosis.2021.12.004. Epub 2021 Dec 12. PMID 34922192
- [Derived] Jacobi N, Walther C, Borof K, Heydecke G, Seedorf U, Lamprecht R, Beikler T, Debus SE, Waldeyer C, Blankenberg S, Schnabel RB, Aarabi G, Behrendt CA. The Association of Periodontitis and Peripheral Arterial Occlusive Disease in a Prospective Population-Based Cross-Sectional Cohort Study. J Clin Med. 2021 May 11;10(10):2048. doi: 10.3390/jcm10102048. PMID 34064657